CLINICAL TRIAL: NCT06454656
Title: A "MOtor Learning Based Intervention for Lower Extremities (MOBILE)" to Target Walking Performance in Ambulant Children With Cerebral Palsy: A Feasibility Study
Brief Title: A Motor Learning Intervention to Target Walking Performance in Ambulant Children With Cerebral Palsy
Acronym: MOBILE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Principal Investigator, Catriona O'Shaughnessy, Professional Doctorate Scholar, Royal College of Surgeons, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-163
Record Dates: First submitted 2024-05-24; First posted 2024-06-12 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy; Walking, Difficulty; Spastic Diplegia; Hemiplegic Cerebral Palsy
Keywords: Motor Learning Theory; Neuroplasticity; Neurological Rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants will undergo 30 hours of therapy over 6 weeks in format of their choosing.
  A minimum of 24 hours must be completed in clinic with the rest made up of home program.
  Interventions: Other: MOBILE

INTERVENTIONS:
Other: MOBILE — Intensive motor learning based intervention to target specific walking goals as identified using the Gait Outcome Assessment List.
  Full Protocol outlining strategies available on request.
  Three key principles underpin the intervention:
  Principle 1: The type of task
  Principle 2: The type of practice
  Principle 3: The type of Feedback
  Other Names: MOtor learning Based Intervention for Lower Extremities

SUMMARY:
The goal of this clinical trial is to learn if a new therapy approach to improve walking ability in children with Cerebral Palsy is acceptable to the children and the families in a community setting.

The main questions we look to answer are:

1. Do the children/teens tolerate the therapy and feel that it is helpful?
2. Do the parents/ families feel the therapy helps and is easy to commit to?
3. Do the children/teens complete all their therapy sessions and assessments as planned?

The participants will trial the therapy for 30 hours over 6 weeks and will perform assessments before and after to see if they meet their goals. They will also be interviewed to see how they felt about the therapy when they finish.

DETAILED DESCRIPTION:
The therapy being trialed in this study uses motor learning theory to try and improve or change walking patterns to improve the child/teen's walking goal.

Therapy will target their own walking goal and they can choose the format of their therapy as long as they complete 30 hours of which 24 hours must be in the clinic within a 6 week period.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Cerebral Palsy (GMFCS Levels I-III)
* Has a specific walking related goal
* Has capacity to follow instruction
* Has a primary caregiver who can support a home program

Exclusion Criteria:

* Has had surgery within 6 months of intervention start date
* Has had botox/ baclofen within 3 months of intervention start date
* Has a dual diagnosis that impacts ability to follow instruction
* Has a significant cognitive impairment

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | rolling recruitment over 1.5 years
  Percentage of eligible numbers recruited
Adherence to Intervention | Duration of study 2 years
  Percentage of total hours practiced/ planned dose (30 hours)
Retention | Duration of study 2 years
  Percentage of recruited participants at final follow up
Adverse Events | Duration of study 2 years
  Measured as Yes or No with description
Fidelity to Intervention Protocol | Duration of study 2 years
  Checklist to measure extent of motor learning principles included in sessions
Feasibility of Outcome Measures (Participant) | Duration of study 2 years
  Participant experience of outcomes captured by semi-structured interviews.
Feasibility of Outcome Measures (Assessor) | Duration of study 2 years
  Assessor experience of outcomes captured by semi-structured interview.
Acceptability of Intervention | Duration of study 2 years
  Semi-structured interviews of participants and parents to capture acceptability of intervention using Framework of acceptability
Time taken to complete Outcome Measures | Duration of study 2 years
  Measured in Minutes

SECONDARY OUTCOMES:
Gait Outcome Assessment List | baseline, upon completion of intervention (2-6 weeks) and 3 month follow up, rolling through duration of study 2 years
  parent/self-report questionnaire developed to measure functional mobility and goals for ambulant children with CP. This measure will be used to power a future definitive trial.
6 minute walk test | baseline, upon completion of intervention (2-6 weeks) and 3 month follow up, rolling through duration of study 2 years
  This is a measure of gait endurance and has been validated for use in CP. Gait speed will also be calculated using this measure.
10 meter self-selected walking speed | baseline, upon completion of intervention (2-6 weeks) and 3 month follow up, rolling through duration of study 2 years
  habitual walking speed selected as it correlates well with habitual physical activities.
Modified timed up and go | baseline, upon completion of intervention (2-6 weeks) and 3 month follow up, rolling through duration of study 2 years
  tests balance and basic mobility in children with physical disabilities and has been validated for use in CP
ankle and knee Range of motion | baseline, upon completion of intervention (2-6 weeks) and 3 month follow up, rolling through duration of study 2 years
  CPIP measures of ankle DF and popliteal angle
Child Health Utilities Index CHU-9D | baseline, upon completion of intervention (2-6 weeks) and 3 month follow up, rolling through duration of study 2 years
  self-report measure that can calculate quality adjusted life years to measure quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ailish Malone, PHD, Principal Investigator — Royal College of Surgeons
Locations (1):
- Enable Ireland Bangla Therapy Centre, Balrath, Meath, Ireland